CLINICAL TRIAL: NCT05894369
Title: Influence Mechanism of Tumor Microenvironment Changes on Neoadjuvant Therapy for Esophageal Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Yongshun Chen, professor, Renmin Hospital of Wuhan University
Other Study IDs: WDRY2023-K056
Record Dates: First submitted 2023-05-26; First posted 2023-06-08 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Cancer
Keywords: neoadjuvant therapy; immunotherapy; overall survival; efficacy; safety
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neoadjuvant chemotherapy combi

SUMMARY:
To evaluate the predictive value and mechanism of inflammatory factors in peripheral blood on the prognosis of patients, and to explore the influencing factors of inflammation and tumor microenvironment on the efficacy of neoadjuvant chemotherapy combined with immunotherapy for esophageal cancer. To explore the predictors of neoadjuvant therapy in patients with esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Patients with esophageal cancer admitted to Hubei Provincial People's Hospital from May 2023 to December 2024 were collected (the estimated number of patients included is 60). Collect research objects: 1. Baseline information: gender, age, tumor location, T stage, N stage, and BMI, etc. The tumor staging and grading are determined according to the eighth edition of American Joint Committee on Cancer esophageal cancer staging; 2. Laboratory data; Blood routine, liver and kidney function, electrolyte, coagulation function, tumor markers and cytokines were collected before neoadjuvant chemotherapy combined with immunotherapy, after 2 cycles of treatment and after 4 cycles of treatment (if applicable). After every two cycles of treatment, the remission status of the disease was evaluated by CT or gastroscopy in the routine treatment. To evaluate the predictive value and mechanism of peripheral blood inflammatory factors on the prognosis of patients, and to explore the influencing factors of inflammation and tumor microenvironment on the efficacy of neoadjuvant chemotherapy combined with immunotherapy for esophageal cancer.

ELIGIBILITY:
Inclusion criteria：

The patient's age between 18 to 80 years old; Esophageal squamous cell carcinoma with definite pathological diagnosis and II-IVA clinical stage Preoperative neoadjuvant chemotherapy combined with immunotherapy The score of eastern cooperative oncology group is 0 ~ 1 Exclusion criteria

The estimated survival time is less than 6 months; The first diagnosis had distant metastasis Suffering from malignant tumor or accompanying malignant disease in the past 5 years Pregnant or pregnant women. Vulnerable groups (those without informed ability, minors, vagrants, students and subordinates of researchers, employees of bidders)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Tumor diameter | 1 year
  The tumor diameter will be measured to evaluate the therapeutic effect

SECONDARY OUTCOMES:
Overall survival | 1 year
  The survival time of patients is calculated from first treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin hosptial of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
This study is prospective, so it is limited by some uncertainties.